CLINICAL TRIAL: NCT05248425
Title: A Randomized Study to Measure and Enhance the Health Related Quality Of Life in Cancer Patients Receiving Immune Checkpoint Modulators
Brief Title: Study to Measure and Enhance the Health Related Quality Of Life in Cancer Patients
Acronym: ME-Q
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Dacima Software Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-6057
Record Dates: First submitted 2022-02-11; First posted 2022-02-21 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Cancer
Keywords: ICMs; Immune Checkpoint Modulators
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): All participants will answer questionnaires at specified time points. This arm will receive usual care and their questionnaire responses will not be reviewed.
- Monitored (Experimental): All participants will answer questionnaires at specified time points. The monitored arm will have their responses reviewed for new or worsening symptoms which will be assessed and managed by a study nurse in addition to usual care.
  Interventions: Other: Nurse Monitoring

INTERVENTIONS:
Other: Nurse Monitoring — Questionnaire responses that indicate new or worsening symptoms will be monitored by a study nurse who will contact the participant for clinical assessment and develop a management plan following irAEs management guidelines.
  Arms: Monitored

SUMMARY:
The ME-Q study aims to validate a patient reported outcome tool called FACT-ICM, which measures health related quality of life (HRQOL) in patients receiving immune checkpoint modulator (ICM) therapy. In addition, this trial seeks to answer if HRQOL can be improved by monitoring and managing patient symptoms whilst they are treated with ICMs.

DETAILED DESCRIPTION:
Immunotherapy has revolutionized cancer care by extending survival, but with a unique set of toxicities known as immune-related adverse events (irAEs), less is known about impact of ICMs on HRQOL.

The ME-Q trial will produce two major innovations: 1) the first validated tool to measure HRQOL in patients on ICMs that can be used in clinical trials and routine clinical care; and 2) a system to monitor and manage patient symptoms on ICMs which can enhance health care delivery for these cancer patients.

ME-Q will randomize patients who are treated with standard of care ICMs to either a monitoring arm developed specifically for this trial or the usual care arm, which is currently how they are managed. All participants will respond to HRQOL questionnaires of which FACT-ICM is a core component. A study nurse will review and manage responses which indicate new or worsening symptoms for those in the monitoring arm. The nurse will contact the patient via telephone or video teleconferencing to conduct a clinical assessment and develop a management plan following irAEs management guidelines. We hypothesize that patients on the monitoring arm will have better HRQOL, longer overall survival, fewer presentations to the emergency department and less hospital admissions than the usual care arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosed with advanced, incurable solid tumors
* Eligible for immunotherapy (monotherapy or combination ICM)
* Life expectancy ≥ 6 months
* ECOG PS 0-3
* Fluent in English
* Able to provide informed consent
* Able to complete questionnaires using digital device or web based application

Exclusion Criteria:

* Participation in a therapeutic clinical trial testing anticancer therapies
* Receiving adjuvant immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Health Related Quality Of Life measured via Functional Assessment of Cancer Therapy - General (FACT-G) at 4 months from baseline, lower scores meaning worse outcome | Baseline; 4 months

SECONDARY OUTCOMES:
Validity testing of FACT-ICM using Pearson or Spearman correlations between toxicity subscale and FACT-G components of the FACT-ICM and FACT-G scores | Baseline; Up to 45 months
  Test-retest reliability, discriminative capacity, construct validity, responsiveness and minimally clinically important differences of FACT-ICM subscale
Overall survival at 1 year and 2 years | 1 year; 2 years
Evaluate quality adjusted survival | Baseline; Up to 45 months
  Average FACT-G scores will be multiplied by survival times for each reporting interval, with values summed to yield a total number of quality adjusted life months
Time to first Emergency Department visit and time to first hospitalization | Up to 45 months
Time on ICM therapy and time to subsequent therapy | Up to 45 months
Adherence rate and completion rate of FACT-ICM | Up to 45 months
  Ratio of completed ePRO/ratio of ePRO reports that should have been completed within 72 hours of email alert

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Hansen, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada